CLINICAL TRIAL: NCT01819207
Title: Evaluation of the Coagulation Profile by Thromboelastography in Bariatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1492MF
Record Dates: First submitted 2013-03-24; First posted 2013-03-27 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2013-03

CONDITIONS: Bariatric Patients Undergoing Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TEG group (Experimental)
  Interventions: Other: blood test by thromboelastography

INTERVENTIONS:
Other: blood test by thromboelastography

SUMMARY:
thromboelastography can identify alteration in the coagulation profile in bariatric patients who undergo sleeve gastrectomy or gastric bypass

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing bariatric surgery

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
coagulation profile by thromboelastography | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Naharia Medical Center, Nahariya, Israel

REFERENCES:
- [Background] Munro TG. Glass is detectable on plain radiographs. CMAJ. 1989 Feb 15;140(4):365. No abstract available. PMID 2914257